CLINICAL TRIAL: NCT03674619
Title: A Randomised Controlled Trial Comparing the Effectiveness of Surgical and Nonsurgical Treatment for Cervical Radiculopathy
Brief Title: Cervical Radiculopathy Trial
Acronym: CRT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mirad Taso, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017/2125
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Active Comparator): Anterior discectomy
  Interventions: Procedure: Anterior discectomy
- Conservative treatment (Active Comparator): Patients will attend an experienced specialist in physical medicine and rehabilitation and a physiotherapist.
  Interventions: Behavioral: Conservative treatment

INTERVENTIONS:
Procedure: Anterior discectomy — Anterior discectomy will be performed and a microscope is used. After separation of the platysma muscle the pre-vertebral space is reached by an approach medial to the sternocleido-mastoid muscle and the carotid artery and lateral to the trachea and oesophagus. Then the disc is incided and the corpora are distracted to perform discectomy. Usually the posterior ligament is cut and the spinal root is decompressed and if necessary the arthritic rims are removed. An inter-vertebral fusion device is inserted, two levels are allowed in the spondylosis study.
  Arms: Surgical treatment
Behavioral: Conservative treatment — Patients will first attend an experienced specialist in physical medicine and rehabilitation who will answer concerns and questions and if necessary repeat the information given before inclusion. The aim of the brief intervention is to promote better understanding and coping of the condition. The intervention will include supervision by a physiotherapist (6 sessions altogether) and provide advice on how to handle secondary neck muscle pain and dysfunction, reduce eventual fear avoidance, and advice to stay active.
  Arms: Conservative treatment

SUMMARY:
The primary aim of the present project is to compare the effectiveness of surgery and nonsurgical treatment in patients with cervical radiculopathy caused by either disc herniation or spondylosis. Secondary aims are to evaluate cost-effectiveness and predicting factors of success of the two treatments, and to explore the terms success rate and expectations by asking the patients to fill in their expected primary outcome score at baseline.

DETAILED DESCRIPTION:
Cervical radiculopathy is usually caused by disc herniation or spondylosis. Prognosis is expected to be good in most patients but there is limited scientific evidence about the indication for non-surgical and surgical treatment.

Two randomised controlled trials comparing cervical decompression and non-operative treatment with cost-effectiveness analysis and assessment of expectations and predictors of outcome. The main research question will be evaluated at one-year follow-up.

1. To test the hypothesis that the effectiveness of surgery as measured by the change in Neck Disability Index (NDI) at 1-year follow-up in patients with cervical radiculopathy is not different from non-surgical treatment in:

   1. Study 1: one level disc herniation (C5/6 or C6/7)
   2. Study 2: one or two level spondylosis (C5/6 and/or C6/7)
2. To test the hypothesis that surgery is more effective in patients with more clinical finding (dermatomal sensory loss, myotonal weakness and reflex disturbance) at baseline when adjusted for other possible predictors such as age, gender, baseline pain, duration, radiological findings, expectations, and psychological factors).
3. To estimate cost-effectiveness for health care costs and societal costs (including sickness absence) in surgical versus non-surgical patients.
4. To assess radiological (MRI and CT) measurements of foraminal area and nerve compression and if changes can predict clinical changes (NDI and arm pain) at 1-year .
5. To evaluate treatment outcome expectations at baseline asking the patients to fill in their expected improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65 years.
* Study 1: Neck and arm pain for at least 3 months with a corresponding herniation involving one cervical nerve root (C6 or C7) Study 2: Neck and arm pain for at least 3 months with a corresponding spondylosis involving C6 and/or C7) .
* Pain intensity of arm pain of at least 4 on a scale from 0 (no pain) to 10 (worst possible pain)
* Willing to accept either of the treatment alternatives
* NDI > 30

Exclusion Criteria:

* Patients with any previous cervical fractures or cervical spine surgery;
* Signs of myelopathy;
* Rapidly progressive paresis or paresis < grade 4;
* Pregnancy;
* Arthritis involving the cervical spine;
* Infection or active cancer;
* Generalised pain syndrome;
* Serious psychiatric or somatic disease that exclude one of the treatment alternatives;
* Concomitant shoulder disorders that may interfere with outcome;
* Abuse of medication/narcotics,
* Not able to understand written Norwegian,
* Not willing to accept one of the treatment alternatives.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Follow-up at 52 weeks is the primary end point.
  Consists of ten questions about pain related disability and include items such as by example headache, concentration, reading and sleep. Each item is rated by choosing one of five response categories and transformed to a total score from 0 to 100 (worst possible). The Norwegian version has been validated in patients with neck pain and with cervical radiculopathy.

SECONDARY OUTCOMES:
Neck pain | 52 weeks
  Neck pain measured by Numeric Rating Scale (NRS) from 0 (no pain to 10 (worst imaginable pain).
EuroQol (EQ-5D-5L and EQ-VAS) | 52 weeks
  EQ-5D-5L includes five domains: mobility; self-care, daily activities, pain/discomfort, and anxiety/depression and each has three response categories. The responses are transformed into and index to value the patients' health related quality of life for the cost utility analyses. Patients score their health from 0 (as bad as possible) to 100 (best possible) by EQ-VAS. The Norwegian version has been validated in patients with back pain, idiopathic scoliosis, and cervical radiculopathy.
Fear-avoidance beliefs | 52 weeks
  Evaluated with the Fear Avoidance Beliefs Questionnaire
Emotional distress | 52 weeks
  Assessed by the 10-question version of the Hopkins Symptom Check List
Perceived recovery | 52 weeks
  Perceived recovery or change of the main symptom rated on a numeric scale ranging from -9 (worst possible change) to 9 (best possible change)
Sickness absence data | 52 weeks
  Sickness absence data will be collected from the National Social Security Institution for the year before and after inclusion.
Dysphagia | 52 weeks
  As recorded by The Dysphagia Short Questionnaire
Medicine consumption | 52 weeks
  Questions related to pain medication usage.
Patient expectations | At inclusion
  Exploring patient expectations ahead of treatment. The patients are asked to fill out the Neck Disability Index pretending they are at 52 weeks post treatment and selecting the lowest category they would be content with for each item. The patients are also asked to report what they expect their symptoms to be like 52 weeks ahead (ranging from much worse to much better), registered for arm pain, neck pain and headache separately.
Success rate | 52 weeks
  Exploring global success rate by asking the patients about how the arm pain and neck pain is compared to prior to treatment (ranging from much worse to much better).
Arm pain | 52 weeks
  Arm pain measured by Numeric Rating Scale (NRS) from 0 (no pain to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ivar Brox, MD PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Taso M, Sommernes JH, Sundseth J, Pripp AH, Bjorland S, Engebretsen KB, Kolstad F, Zwart JA, Brox JI. Surgical versus Nonsurgical Treatment for Cervical Radiculopathy. NEJM Evid. 2025 Apr;4(4):EVIDoa2400404. doi: 10.1056/EVIDoa2400404. Epub 2025 Mar 25. PMID 40130970
- [Derived] Taso M, Sommernes JH, Bjorland S, Zwart JA, Engebretsen KB, Sundseth J, Pripp AH, Kolstad F, Brox JI. What is success of treatment? Expected outcome scores in cervical radiculopathy patients were much higher than the previously reported cut-off values for success. Eur Spine J. 2022 Oct;31(10):2761-2768. doi: 10.1007/s00586-022-07234-7. Epub 2022 May 13. PMID 35551484
- [Derived] Taso M, Sommernes JH, Kolstad F, Sundseth J, Bjorland S, Pripp AH, Zwart JA, Brox JI. A randomised controlled trial comparing the effectiveness of surgical and nonsurgical treatment for cervical radiculopathy. BMC Musculoskelet Disord. 2020 Mar 16;21(1):171. doi: 10.1186/s12891-020-3188-6. PMID 32178655

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT03674619/Prot_SAP_003.pdf